CLINICAL TRIAL: NCT05112718
Title: The Use of Platelet Rich Plasma (PRP) as a Treatment of the Female Stress Urinary Incontinence
Brief Title: Platelet Rich Plasma in Women With Urinary Incontinence
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Themos Grigoriadis, Associate Professor of Gynecology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 420/20-09-2019
Record Dates: First submitted 2021-10-26; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Urinary Incontinence; Stress Urinary Incontinence
Keywords: incontinence; urinary incontinence; stress urinary incontinence; platelet rich plasma; PRP,; outpatient treatment; nonsurgical treatment
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma (Experimental): The patients who receive PRP injections
  Interventions: Biological: Platelet Rich Plasma Injections
- Normal Saline (Sham Comparator): The patients who receive normal saline
  Interventions: Other: Normal Saline Injections

INTERVENTIONS:
Biological: Platelet Rich Plasma Injections — PRP injected into 9 sites of the distal anterior one-third of the vagina using a small 30-gauge needle. The injections were performed at 10, 12 and 2 o'clock in 3 different levels of the urethra 1-2 cm apart (distal, mid and proximal).
  The participants will receive 2 PRP injections at 4-6-week intervals. Xylocaine gel 2% is applied to the distal anterior vaginal wall 20 minutes before injections.
  Arms: Platelet Rich Plasma
Other: Normal Saline Injections — Normal saline injected into 9 sites of the distal anterior one-third of the vagina using a small 30-gauge needle. The injections were performed at 10, 12 and 2 o'clock in 3 different levels of the urethra 1-2 cm apart (distal, mid and proximal).
  The participants will receive 2 injections at 4-6-week intervals.
  Arms: Normal Saline

SUMMARY:
Stress urinary incontinence (SUI) is defined as involuntary loss of urine on effort or physical exertion or on sneezing or coughing. Platelet-rich plasma (PRP) is an autologous solution of human plasma containing various growth factors witch enhance regeneration and healing process. The aim of this study is to evaluate the efficacy and safety of PRP in the treatment of the female SUI.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with stress urinary incontinence

Exclusion Criteria:

* pregnancy,
* history of active malignant pathology,
* mental disorders making them unable to give consent,
* undiagnosed abnormal uterine bleeding,
* genitourinary fistula,
* anti-incontinence surgery,
* pelvic organ prolapse stage > 2 according to POP-Q system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Stress urinary incontinence symptoms | 6-12 months
  International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) Number of items: 12
  Question items:
  Nocturia,Urgency, Bladder pain, Frequency, Hesitancy, Straining, Intermittency, Urge urinary incontinence, Frequency of urinary incontinence, Stress urinary incontinence, Unexplained urinary incontinence, Nocturnal enuresis
  Completion time: 4-5 minutes
  Scoring:
  0-16 filling symptoms subscale 0-12 voiding symptoms subscale 0-20 incontinence symptoms subscale 0-48 where all subscale scores are added. Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient
  Higher scores indicate greater impact of individual symptoms for the patient.

SECONDARY OUTCOMES:
Impact of urinary incontinence on the quality of life | 6-12 months
  King's Health Questionnaire (KHQ)
  Description: The KHQ is an assessment of health-related quality of life related to a specific condition.
  Format: 21 items about urinary tract symptoms yield scores in 9 domains (general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy & severity of symptoms).
  Scoring: Each item is rated using a 4 or 5 points likert scale. Domain scores range from 0 (best) to 100 (worst). There are 2 single-item domains (general health perceptions, and incontinence impact) and the severity of symptoms domain is scored using a scale from 0 (best) to 30 (worst).
Assessment of urine loss (1-hr pad test) | 6-12 months
  One-hour pad test standardized by International Continence Society (ICS):
  * started by putting one pre-weighted pad,
  * patient drinks 500 ml in <15 min- then sits or rests,
  * patient walks for 30 min,
  * patient performs the following activities: standing up from sitting, coughing vigorously, running on the spot for 1 min, bending to pick up an object from the floor, and washing hands in running water for 1min
  * the total amount of urine leaked is determined by weighing the pad.
  Interpretation:
  The upper limit of weight increase for the 1-hr test in continent women is 1.4 grams.
  A weight gain of less than 1.4 g during 1-hr test could be a result of sweating or vaginal discharge.
  An increase of 1-10 g is classified as representing mild incontinence, 11-50 g moderate and >50 g severe incontinence.
Level of discomfort during injections (VAS score) | 6-12 months
  The visual analog scale (VAS) is pain rating scale. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Patient Global Impression of Improvement | 6-12 months
  The Patient Global Impression of Improvement (PGI-I) is a validated generic tool for assessment of the over-all improvement or deterioration that the patient may experience following the treatment.
  The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1. Very much better to 7. Very much worse.
  Therefore, lower values correlate with increased satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Athanasiou, Professor, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Urogynecological Unit of Alexandra Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawood AS, Salem HA. Current clinical applications of platelet-rich plasma in various gynecological disorders: An appraisal of theory and practice. Clin Exp Reprod Med. 2018 Jun;45(2):67-74. doi: 10.5653/cerm.2018.45.2.67. Epub 2018 Jun 29. PMID 29984206
- [Background] Alves R, Grimalt R. A Review of Platelet-Rich Plasma: History, Biology, Mechanism of Action, and Classification. Skin Appendage Disord. 2018 Jan;4(1):18-24. doi: 10.1159/000477353. Epub 2017 Jul 6. PMID 29457008
- [Background] Schreiber Pedersen L, Lose G, Hoybye MT, Elsner S, Waldmann A, Rudnicki M. Prevalence of urinary incontinence among women and analysis of potential risk factors in Germany and Denmark. Acta Obstet Gynecol Scand. 2017 Aug;96(8):939-948. doi: 10.1111/aogs.13149. Epub 2017 May 20. PMID 28401541
- [Background] Behnia-Willison F, Nguyen TTT, Norbury AJ, Mohamadi B, Salvatore S, Lam A. Promising impact of platelet rich plasma and carbon dioxide laser for stress urinary incontinence. Eur J Obstet Gynecol Reprod Biol X. 2019 Oct 22;5:100099. doi: 10.1016/j.eurox.2019.100099. eCollection 2020 Jan. PMID 32021973
- [Derived] Grigoriadis T, Kalantzis C, Zacharakis D, Kathopoulis N, Prodromidou A, Xadzilia S, Athanasiou S. Platelet-Rich Plasma for the Treatment of Stress Urinary Incontinence-A Randomized Trial. Urogynecology (Phila). 2024 Jan 1;30(1):42-49. doi: 10.1097/SPV.0000000000001378. Epub 2023 Jun 1. PMID 37493287